CLINICAL TRIAL: NCT00517335
Title: The Evaluation of Brain Neuronal Activity in Response to Natural (Sucrose) and Artificial (Sucralose) Taste Stimuli- Does Caloric Content Matter to the Brain?
Brief Title: Evaluating the Brain's Response to Natural Versus Artificial Sweetener in Women Who Have Had an Eating Disorder
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Walter Kaye, MD Professor of Psychiatry, University of California San Diego
Other Study IDs: R01MH046001 (NIH); R01MH046001 (NIH); DATR A3-NSS
Record Dates: First submitted 2007-08-14; First posted 2007-08-16 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2015-04

CONDITIONS: Eating Disorders
Keywords: anorexia nervosa; bulimia nervosa
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Bulimia Nervosa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — If desired subjects have a chance to be a part of a DNA blood draw aspect of the study

GROUPS / COHORTS (3):
- 1: Women who are healthy controls
  Interventions: Procedure: Functional magnetic resonance imaging (fMRI) scan
- 2: Women who have recovered from bulimia
  Interventions: Procedure: Functional magnetic resonance imaging (fMRI) scan
- 3: Women who have recovered from anorexia
  Interventions: Procedure: Functional magnetic resonance imaging (fMRI) scan

INTERVENTIONS:
Procedure: Functional magnetic resonance imaging (fMRI) scan — Healthy control women, recovered bulimia women, and also recovered anorexia women will complete specific tasks in an fMRI scanner that will take up to 60 minutes.
  Other Names: Neurobiology of Eating Disorders; fMRI imaging of Anorexia and Bulimia Nervosa

SUMMARY:
This study will compare the brain's ability to distinguish between natural and artificial sweeteners in women with and without a history of eating disorders.

DETAILED DESCRIPTION:
Eating disorders often result in serious illness and can lead to prolonged health complications, including heart and kidney problems, digestive disorders, nerve damage, and low blood pressure. Anorexia nervosa and bulimia nervosa are examples eating disorders. People with anorexia nervosa do not eat enough in fear of becoming overweight, resulting in extreme weight loss. People with bulimia nervosa first binge by consuming hundreds or even thousands of calories within a very short time period and then purge by either vomiting or using laxatives. Women are at a greater risk of developing the disorders, particularly when they are between the ages of 12 and 24. Treatments for eating disorders typically include nutrition counseling, psychotherapy, and medication. To better understand eating disorders, this study will compare the brain's ability to distinguish between natural and artificial sweeteners in women with and without a history of eating disorders.

All participants in this observational study will be administered a taste test to determine if they can consciously differentiate between a sugar solution and an artificially sweetened solution. Participants may also perform several brief computerized tests, ranging from 3 to 10 minutes each, to evaluate thinking, memory, and information processing skills. Participants who cannot tell the difference between the solutions will undergo a functional magnetic resonance imaging (fMRI) scan, which will take pictures of the brain and blood flowing through the brain. Prior to the scan, blood and urine collection may occur, and participants may complete two additional computerized tests. The scan will require 60 to 90 minutes to complete. During the scan, participants will hold two thin tubes in their mouth. At various intervals, these tubes will deliver 1 ml of liquid containing either sugar water or an artificial sweetener into each participant's mouth. A screen projection of abstract pictures will also be shown to each participant throughout the scan, either before the liquid is delivered or alone. This study will require a 6- to 9-hour time commitment. The results from this study may provide valuable information regarding anorexia nervosa and bulimia nervosa and may eventually lead to the development of new and better treatment options for these complex and serious disorders.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed
* Recovered from anorexia or bulimia nervosa at least 12 months prior to study entry
* Met DSM criteria for anorexia or bulimia nervosa at one time within 3 years prior to study entry

Exclusion Criteria:

* Pregnant or breastfeeding
* Currently taking any medication (except birth control)
* Any current mental illness
* Any metal in body

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will include women between the ages of 18 and 45 who have recovered from anorexia or bulimia nervosa for over 1 year and have no current medical problems.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2005-05; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Watler Kaye, MD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Eating Disorders Treatment and Research Center, La Jolla, California, United States